CLINICAL TRIAL: NCT03561272
Title: The Validation of a Novel Adherence Method for Oral Oncolytics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2015.030; HUM00098103 (Other: University of Michigan)
Record Dates: First submitted 2018-03-02; First posted 2018-06-19 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Patient Reported Adherence (No Intervention): Adherence assessment via phone call or in person
- Smart Phone Application (Active Comparator): Adherence assessment via phone app
  Interventions: Other: Smart Phone Application
- POD and Smart Phone Application (Experimental): Adherence assessment via phone app partnered with an automated dispensing machine, a "Pod."
  Interventions: Other: Smart Phone Application; Other: POD

INTERVENTIONS:
Other: Smart Phone Application — Oral medication adherence phone application.
  Arms: POD and Smart Phone Application; Smart Phone Application
Other: POD — Pill dispensing system that dispenses the medication, controls dispensed dosage, and confirms dispensing to patient through wireless communication back to the control center.
  Arms: POD and Smart Phone Application

SUMMARY:
The long-term goal of this research is to apply technologic approaches to improve the use of oral oncolytics. The objective of this study is to assess patient adherence to oral oncolytics and to validate a currently available smart phone application (iRxReminder) partnered with an automated dispensing device, a "Pod", in affecting patient adherence. The rationale for this study is that medication adherence to oncolytics varies and strategies are needed to improve it.

ELIGIBILITY:
Inclusion Criteria:

* Must be > 18 years of age
* Must have a smart phone
* Must be able to have their oral oncolytic filled at the University of Michigan Comprehensive Cancer Center pharmacy and be newly prescribed Capecitabine (Xeloda).

Exclusion Criteria:

* Patients who do not have a smart phone
* Patients who have a serious mental illness or cognitive impairment, e.g., psychosis or dementia.
* Patients who do not speak English
* Patients who cannot fill their oral oncolytic prescription at the University of Michigan Comprehensive Cancer Center Pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
The change in the number of patients that report high adherence over time via smart phone application alone | 0, 4, 8 and 12 weeks
  Adherence will be assessed via smart phone application at baseline, 4, 8 and 12 weeks.
  Adherence reported via the phone application will be done using an adherence question assessment.This assessment is ordinal in nature and asks the patient to rate their adherence on a scale (poor, fair, good, very good, excellent).
The change in the number of patients that report high adherence over time via smart phone application and POD | 0, 4, 8 and 12 weeks
  Adherence will be assessed via smart phone application + POD at baseline, 4, 8 and 12 weeks.
  Adherence reported via the phone application will be done using an adherence question assessment.This assessment is ordinal in nature and asks the patient to rate their adherence on a scale (poor, fair, good, very good, excellent).
  For the Pod there will be continuous adherence assessed via the pod each time the patient administers or does not administer a scheduled dose. This will be figured into the overall adherence rating.
The change in the number of patients that report high adherence over time via telephone/face-to-face visit (self-reported) | 0, 4, 8 and 12 weeks
  Adherence will be assessed via telephone/face-to-face visit (self-reported) at baseline, 4, 8 and 12 weeks.
  Self-reported adherence will be done using an adherence question assessment.This assessment is ordinal in nature and asks the patient to rate their adherence on a scale (poor, fair, good, very good, excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Shawna Kraft, Pharm.D., BCOP, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided